CLINICAL TRIAL: NCT02244229
Title: MICTUS (Multicentre Investigation to Characterise the Effect of Tamsulosin on Urinary Symptoms): A Multicentre, Double-blind, Randomised, Parallel Group Study, Aimed at Characterising the Effect of Tamsulosin, an Uroselective α1- Receptor Blocking Agent, on the Urological Symptoms and Their Impact on General Health Status and Quality of Life in Outpatients Affected by Symptomatic Benign Prostatic Hyperplasia: Comparison With Finasteride.
Brief Title: Study to Evaluate the Therapeutic Action of Tamsulosin and Finasteride in Symptomatic Benign Prostatic Hyperplasia (BPH) Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 527.15
Record Dates: First submitted 2014-09-18; First posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Tamsulosin; Finasteride

ARMS (2):
- Tamsulosin (Experimental)
  Interventions: Drug: Tamsulosin; Drug: Placebo
- Finasteride (Active Comparator)
  Interventions: Drug: Finasteride; Drug: Placebo

INTERVENTIONS:
Drug: Tamsulosin
  Arms: Tamsulosin
Drug: Finasteride
  Arms: Finasteride
Drug: Placebo

SUMMARY:
Study to evaluate the therapeutic effect of tamsulosin and finasteride in symptomatic BPH patients, two medications indicated in BPH belonging to two different pharmacological classes, as evaluated from the point of view of patient's perception of his pathological condition and of the impact of the disease on general health and quality of life

ELIGIBILITY:
Inclusion Criteria:

* Male out-patients aged 50-80 years
* IPSS >= 13 at Visit 1
* Qmax: 4-15 ml/sec at Visit 2
* Residue urinary volume > 400 ml as evaluated by ultrasonography
* SPI >= 7 at Visit 2
* Prostate Specific Antigen (PSA) value < 3 ng/ml at Visit 1, or of 3-10 ng/ml provided that prostate cancer is ruled out on the basis of the usual diagnostic procedures performed at each Centre
* Written informed consent

Exclusion Criteria:

Patients with known history or diagnosis at the time of the screening visit of the following conditions that could influence the end-points of the study:

* Urological disturbances

  * Medical history of pelvic surgery; palpable bladder at the physical examination, or residue urinary volume > 400 ml; known neurological bladder disorder, bladder neck stenosis, urethral stricture, bladder or prostatic cancer, bladder stone, severe diverticulum of the bladder, symptomatic urinary tract infection during the last month, or recurrent urinary tract infections (more than 2 during the last year); hematuria of unknown origin; diseases that may affect micturition (e.g. diabetes mellitus)
* Cardiovascular diseases - The following cardiovascular diseases if occurred in the last 6 months:

  * Myocardial infarction
  * Unstable angina
  * Clinically significant ventricular arrhythmias
  * Heart failure (NYHA classes III/IV)
  * Orthostatic hypotension
  * Cerebral stroke
* Neurological diseases

  * such as senile dementia, multiple sclerosis, Parkinson's disease, psychiatric disturbances, if their severity could have prevented the correct performance of the trial
* Hepatic or renal insufficiency

  * (Biochemistry values 15% outside normal laboratory ranges and regarded as clinically relevant by investigator)
* Clinically significant abnormalities in the results of hematologic and biochemical tests performed on blood samples drawn at the screening visit
* Patients who are taking or have been taking α-blockers for BPH or for hypertension or phytotherapy for BPH in the previous 6 weeks
* Patients who are taking or have been taking finasteride in the last 6 months
* Patients who require concomitant drugs which could influence the pharmacodynamic or pharmacokinetic properties of tamsulosin. In particular: alpha-blockers and mixed alpha-beta blockers, alpha- agonists, anti-cholinergics
* Patient who are or have been taking part in a clinical study in the previous 3 months
* Patients who have hypersensitivity or allergic reactions to previously prescribed alpha-blocker(s) or to finasteride
* Patients judged by the investigator to be inappropriate for inclusion in the study

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 403 (Actual)
Dates: Start 1998-04; Primary Completion 2000-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Symptom Problem Index (SPI) by means of validated patient questionnaire | Baseline, after 26 weeks of treatment

SECONDARY OUTCOMES:
Change in Symptom Problem Index (SPI) - by means of validated patient questionnaire | up to 52 weeks
Change in International Prostatic Symptom Score (IPSS) | up to 52 weeks
  questionnaire for the self-evaluation of urinary symptoms
Change in Qmax by means of free flow uroflowmetry | up to 52 weeks
Number of patients who withdrew due to inefficacy | up to 52 weeks
Number of patients with adverse events | up to 54 weeks
Number of patients with abnormal changes in laboratory parameters | up to 52 weeks